CLINICAL TRIAL: NCT02168283
Title: Treatment of Asymptomatic Fluid Overload in Peritoneal Dialysis Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Cheuk-Chun SZETO, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BPBCM
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Chronic Kidney Disease; Peritoneal Dialysis
Keywords: cardiovascular disease; hypertension
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- treatment arm (Experimental): active fluid management includes 3 components: dietary counseling, diuretics, and intensive dialysis regimen
  Interventions: Combination Product: treatment arm; Behavioral: Control arm
- control arm (Active Comparator): dietary counseling alone
  Interventions: Behavioral: Control arm

INTERVENTIONS:
Combination Product: treatment arm — Hypertonic peritoneal dialysis cycles
  Arms: treatment arm
Behavioral: Control arm — Dietary counseling

SUMMARY:
INTRODUCTION Peritoneal dialysis (PD) is a life-saving treatment for end-stage renal disease patients. However, cardiovascular disease remains the major cause of morbidity and mortality in PD patients. It is now realized that chronic asymptomatic intravascular hypervolemia is an important cause of cardiovascular disease in PD patients.

OBJECTIVES To determine the effects of treating asymptomatic fluid overload on blood pressure, hospitalization and cardiovascular morbidity in PD patients.

HYPOTHESIS The investigators hypothesize that treating asymptomatic fluid overload could improve the clinical outcome of PD patients.

DESIGN & SUBJECTS This is an open label randomized control trial. The investigators plan to recruit 60 PD patients with asymptomatic fluid overload, defined as overhydration (OH) ≥ 2 liters. Patients will be randomized to active fluid management (treatment arm) or conventional management (control arm).

STUDY INSTRUMENTS Overhydration will be identified by bioimpedance spectroscopy.

INTERVENTIONS For the treatment arm, active fluid management includes dietary counseling, diuretics, and intensive dialysis regimen. For the control arm, patients will only receive dietary counseling. Patients will be followed for one year.

MAIN OUTCOME MEASURES Blood pressure control, number of hospital admission and duration of hospitalization for all cause, and hospitalization for cardiovascular disease during the study period.

DATA ANALYSIS Blood pressure control will be compared by Student's t test. Hospitalization data will be compared by non-parametric Mann Whitney U test.

EXPECTED RESULTS The study will determine the benefit of treating asymptomatic fluid overload in PD patients.

DETAILED DESCRIPTION:
The investigators plan to recruit 60 PD patients with asymptomatic fluid overload, which is defined as overhydration (OH) ≥ 2 liters as measured by bioimpedance spectroscopy. Patients with clinical symptoms of fluid overload (including, but not restricted to, dyspnea on exertion, peripheral edema, pulmonary congestion) will be excluded. The investigators will also exclude patients who are in overt pulmonary edema and required urgent medical care, who have cognitive impairment or problem of communication, unlikely to survive for more than three months, have mechanical problems of the dialysis catheter, or have active peritonitis or peritoneal failure.

ELIGIBILITY:
Inclusion Criteria:

* asymptomatic fluid overload, defined as overhydration (OH) ≥ 2 liters as measured by bioimpedance spectroscopy

Exclusion Criteria:

* clinical symptoms of fluid overload (including, but not restricted to, dyspnea on exertion, peripheral edema, pulmonary congestion)
* overt pulmonary edema and required urgent medical care
* cognitive impairment or problem of communication
* unlikely to survive for more than three months
* mechanical problems of the dialysis catheter
* active peritonitis or peritoneal failure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2017-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
blood pressure control | 1 year
number of antihypertensive medications | 1 year
duration of hospitalization for all cause | 1 year
hospitalization for cardiovascular disease | 1 year

SECONDARY OUTCOMES:
degree of overhydration | 1 year
change in residual GFR | 1 year
nutritional status | 1 year
arterial pulse wave velocity | 1 year
cardiovascular mortality | 1 year
all-cause mortality | 1 year

OTHER OUTCOMES:
cause of hospital admission | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong